CLINICAL TRIAL: NCT04723966
Title: Safety and Efficacy Evaluation of TPN in Preterm Neonates in NICU of Cairo University Children Hospital
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Khalid Mohammed Shehata, doctor, Cairo University
Other Study IDs: MS- 110-2019
Record Dates: First submitted 2021-01-21; First posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: TPN in Preterm

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: TPN — Total parenteral nutrition

SUMMARY:
The aim of this work is evaluation of electrolytes and minerals homeostasis and occurrence of complications among preterm babies receiving total parenteral nutrition, and admitted to the neonatal intensive care units of Cairo University Children hospitals.

ELIGIBILITY:
Inclusion Criteria:

- All preterm infants with gestational age < 34 weeks, Receiving total parenteral nutrition. Normal serum magnesium.

Exclusion Criteria:

* Any full-term neonates Any patient with TORCH infection, chromosomal, metabolic disorders or surgical abnormality of the hepatobiliary system

Ages: 1 Day to 1 Month | Sex: All
Age Groups: Child
Study Population: This study will include all male and female preterm infants receiving total parenteral nutrition in NICU of Cairo university Children hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-04-07 (Actual); Primary Completion 2020-03-07 (Actual); Study Completion 2021-12-07 (Estimated)

PRIMARY OUTCOMES:
electrolyte and mineral disturbance associated with TPN in preterm receiving it | 14 days
  NA, K, MG, P, CA.

SECONDARY OUTCOMES:
prevalence of cholestasis and sepsis in preterm receiving TPN | 14 days
  clinical and laboratory examination

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Cairo, Almanyal, Egypt